CLINICAL TRIAL: NCT04930276
Title: The Impact of Diet-controlled Blood Glucose on Gut Microbiome in Women With Diabetes Mellitus
Brief Title: Diet-glucose-gut Microbiome Net in Women With GDM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: JS-2842
Record Dates: First submitted 2021-04-06; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-04

CONDITIONS: GDM; Blood Glucose; Pregnancy Outcome; Microbiota
Keywords: GDM; diet intervention; microbiome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GDM group (Experimental): After participants are enrolled, they would be given medical nutrient treatment. Besides, they need have a follow-up visit every two weeks. Blood glucose, body weight, lifestyle and clinical information are collected. Blood samples and stool samples are collected in 28 and 32 pregnant weeks, respectively.
  Interventions: Other: Diet intervention
- non-GDM group (Other): After participants enrollment, they also would be given medical nutrient treatment. And the other conditions are same as the group of GDM.
  Interventions: Other: Diet intervention

INTERVENTIONS:
Other: Diet intervention — Professionals will guide participants to have a standard diet and require them to monitor blood glucose by themselves.

SUMMARY:
A prospective cohort study was conducted to :1. explore the effective of diet intervention on blood glucose control; 2. observe the changeable composition of microbiota; 3. seek the possible microbiome intervened to prevent GDM.

DETAILED DESCRIPTION:
1. Gestational diabetes mellitus（GDM） is one of the most complications during pregnancy and it is associated with many adverse outcomes for both mother and children in short or long term. Appropriate nutritional intervention is beneficial for the control of blood glucose. However, the strategy of intervention and mechanism remain uncertain. Previous studies have shown that diet maybe influence blood glucose via effecting the composition of gut microbiome. Recently, most studies collect only one sample and combine with the diet review, which have some limitations in revealing the effect of diet on gut microbiota and the process of change in blood glucose. This study aims to achieve the target of controlling blood glucose via diet intervention, which includes staple food distribution, food list and nutritional advice, describe the change of gut microbiota in women with GDM before and after the intervention via amplicon sequencing, estimate the effectiveness of diet intervention on controlling blood glucose and explore the correlation between the level of blood glucose and transition of bacterial diversity by monitoring blood glucose and glycated hemoglobin. Furthermore, explore the mechanism of "diet-bacterial diversity-blood glucose". Investigators hope deeply understand the mechanism of controlling blood glucose via diet intervention and find the effective diet control, probable bacterial intervention, which may be applied in clinical practice.This project is a prospective cohort study designed to explore the effect of diet to control blood glucose on the composition of gut microbiota in women with GDM.
2. The study aims to enroll 50 participants with GDM and 20 participants with non-GDM. They will be provided with medical nutritional intervention and need to collect stool samples before and after intervention, separately. Nutritional professionals provide nutritional suggestions to manage blood glucose via examining food diary . All participants need exam glycated hemoglobin every two weeks and monitor fast blood glucose and 2 hour postprandial blood glucose in a one day. Total times of monitoring blood glucose is at least three times every week. Researchers record the situation of blood glucose both groups. Besides, participants need collect stool sample at 28 weeks (before the intervention) and 32 weeks (after the intervention), respectively. Samples will be sequenced by amplicon to describe the effects of diet intervention on the gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who can have a regular labor inspection and delivery in the labor inspection hospital;
* The range of age is between 18 to 45 years;
* Pregnancy naturally and singleton pregnancy;
* Pregnant women with or without gestational diabetes diagnosed by oral glucose tolerance test at 24 to 28 weeks of pregnancy;
* Those who can skillfully use social software in mobile phones and obey the plan of follow-ups;
* Those who voluntary signing of informing consent.

Exclusion Criteria:

* Patients with pre-pregnancy diabetes or abnormal oral glucose tolerance test screening in early resulting from high risks or known pre-pregnancy glucose intolerance;
* Those who were estimated by endocrinology that their value of blood glucose is controlled by not only diet interventions but also drugs;
* Pregnant women who used antibiotics before 1 month enrollment ;
* Those who combined some metabolic diseases, such as hematological system diseases and nervous system diseases;
* Those who reject signing inform consent.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
blood glucose | From enrollment to delivery
  Fast blood glucose and glycemic albumin will be combined to evaluate the efficiency of blood glucose control
the composition of gut microbiome | From enrollment to delivery
  the composition of gut microbiome in women with GDM and non-GDM
the glycemic qualification rate | From enrollment to delivery
  the frequency of ideal blood glucose values when participants monitor blood glucose by themselves every during every two weeks

SECONDARY OUTCOMES:
pregnancy outcome | during delivery
  the occurrence of pre-eclampsia , gestational hypertension, macrosomia

CONTACTS AND LOCATIONS:
Overall Officials: Liangkun Ma, Study Chair — Chinese Academic of Medical Science & Peking Union Medical College Hospital
Locations (1):
- Department of ob gyn , Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No